CLINICAL TRIAL: NCT03896516
Title: Manipulating Ghrelin Signaling Via GOAT Inhibition in Alcohol Use Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 999919075; 19-DA-N075
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-03-12

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Problems; Alcohol Craving; Food-Seeking Behaviors; Ghrelin; Ghrelin O-acyltransferase
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GLWL-01, then Placebo (Experimental): Participants receive GLWL-01 450 mg orally twice daily for a minimum of four days (Stage I) followed by a minimum of two day wash-out period then placebo orally twice daily for a minimum of four days (stage II).
  Interventions: Other: Placebo; Drug: GLWL-01
- Placebo, then GLWL-01 (Placebo Comparator): Participants receive placebo orally twice daily for a minimum of four days (Stage I) followed by a minimum of two day wash-out period then GLWL-01 450 mg orally twice daily for a minimum of four days (stage II).
  Interventions: Other: Placebo; Drug: GLWL-01

INTERVENTIONS:
Other: Placebo — Participants receive Placebo orally twice daily.
Drug: GLWL-01 — GLWL-01 is a ghrelin O-acyltransferase (GOAT) inhibitor. Participants receive GLWL-01 orally twice daily.

SUMMARY:
Background:

People with alcohol use disorder (AUD) have trouble controlling their drinking. Medications can help some people with AUD but are not effective for many others. Researchers want to test new drugs to better treat the disease.

Objective:

To see if the investigational drug GLWL-01 is safe to use in people with alcohol problems. Also, to find out if the drug reduces the urge to drink alcohol.

Eligibility:

People ages 18-70 with Alcohol Use Disorder (AUD)

Design:

Participants will be screened under protocol 06-DA-N415.

Participants will be admitted to the inpatient facility, Clinical Research Unit (CRU) on the Johns Hopkins Bayview Medical Center for up to 21 days. They may leave the CRU on specified days pending approval. All their meals will be provided. They cannot drink alcohol.

Participants will take either the study drug or a placebo by mouth twice daily. They will not know which they are receiving.

Participants will complete many questionnaires.

Participants may have urine tests.

Participants will complete tasks on a computer.

Participants will have blood samples obtained on some study days.

Participants will taste and indicate their preference for sweet liquids.

Participants' blood pressure, pulse, respiratory rate, body temperature and weight, heart rate and rhythm will be measured.

Participants will have breath testing to obtain information about smoking.

Participants will be exposed to alcohol cues, water, and food cues in a bar-like room. Cues are things that might make them feel the urge to eat or drink alcohol.

Participants will take part in a virtual buffet experiment - They will wear a virtual reality headset, walk around a virtual room, and select virtual food and drink.

DETAILED DESCRIPTION:
Background and Objective: Acyl-ghrelin is a 28-amino acid peptide that stimulates appetite and food intake. It is an endogenous ligand for the growth hormone secretagogue receptor (GHS-R1a). Preclinical studies suggest that acyl-ghrelin increases alcohol intake and decreases in acyl-ghrelin and GHS-R1a function suppresses alcohol consumption. Furthermore, previous human studies indicate a positive correlation between endogenous ghrelin levels and alcohol craving and drinking. In clinical studies conducted by our group with individuals with AUD, intravenous (IV) acyl-ghrelin administration, versus placebo 1) increased alcohol craving during alcohol cue-exposure and 2) increased IV alcohol self-administration as well as decreased latency to first infusion of alcohol and 3) increased brain activation in the amygdala in anticipation of alcohol reward.

Together, this preclinical and human data suggest that manipulating the ghrelin signal may be a novel and potentially effective pharmacological approach to treat individuals with alcohol use disorder.

After the discoveries of GHS-R1a and acyl-ghrelin, a next step was identifying ghrelin O-acyltransferase (GOAT) the enzyme that catalyzes the conversion of des-acyl-ghrelin (DAG) to acyl-ghrelin via octanoylation. GOAT is thus the master switch for the ghrelin system , as acyl-ghrelin, not DAG, is biologically active at the GHSR-1a. GOAT s structure is highly conserved, is produced by endocrine cells in the stomach and is co-expressed with ghrelin. Therefore, GOAT is a promising target for manipulating the ghrelin system by altering the peripheral acyl-to-total ghrelin ratio (where total ghrelin = acyl-ghrelin + DAG). Recently, the ghrelin system has been investigated as a potential treatment target for AUDs.

As such, an oral bioavailable GOAT inhibitor offers encouraging potential as a treatment for alcohol use disorder. GLWL-01 is an existing GOAT inhibitor for which GLWL Research Inc. has recently and successfully completed a first-in-human safety clinical trial. The goal of this protocol is to conduct a proof-of-concept human laboratory study to assess a potential early signal of efficacy of GLWL-01 in relation to alcohol-related outcomes.

Study population: Males and females (N = 43) with alcohol use disorder.

Study Design: A within-subject, counterbalanced, double-blind, placebo-controlled study. Participants will take GLWL-01 450 mg b.i.d. or matched placebo for a minimum of 4 days (Stage I). After a minimum 2 day wash-out window, Stage II will take place during which the counterbalanced study drug will be administered for a minimum of 4 days.

Primary outcome measure: The co-primary aims will be to determine whether: 1) the number of adverse events (AEs) experienced differ in the GLWL-01 condition, compared to placebo; and 2) GLWL-01, compared to placebo, reduces alcohol cue-elicited craving using a validated alcohol cue-reactivity procedure.

Secondary outcome measures: The main secondary aim will be the effects of GLWL-01 on food choices using a virtual buffet experimental procedure. We will also monitor a wide range of behavioral measures including e.g., pain, anxiety, depression, alcohol craving and withdrawal, and smoking.

ELIGIBILITY:
INCLUSION CRITERIA:

* Alcohol Use Disorder (Minimum 2 symptoms on a validated diagnostic tool e.g., the Mini-International Neuropsychiatric Interview (MINI) or the Structured Clinical Interview for DSM Disorders (SCID)
* Male or female individuals 18-70 years old (inclusive)
* Able to speak, read, write and understand English
* Most recent urine drug test for benzodiazepines, barbiturates, cocaine metabolites, morphine, oxycodone, methadone, amphetamine, & buprenorphine is negative.
* Most recent Clinical Institute Withdrawal Assessment for Alcohol - revised (CIWA-Ar) score is less than or equal to 8

Males only:

-Males agrees agree to sexual abstinence or to use a reliable method of birth control during the study and three months following the last dose of the study drug. Acceptable methods of birth control may include: 1) condom with spermicide; 2) diaphragm with spermicide; or 3) female condom with spermicide.

Females only:

-Women of child-bearing potential may participate in the study:

* if they test negative for pregnancy (based on a urine pregnancy test) prior to initiation of treatment
* they must also agree to use either one highly effective method of contraception or a combination of two effective methods of contraception during the study.

  * Highly effective method may include hormonal contraceptives (e.g., combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device or/ intrauterine system; vasectomy and tubal ligation.
  * Effective methods may include barrier methods of contraception (e.g., male condom, female condom, cervical cap, diaphragm, contraceptive sponge)

Women may choose to use a double-barrier method of contraception. Barrier methods without concomitant use of a spermicide are not reliable or an acceptable method. Thus, each barrier method must include use of a spermicide. It should be noted that the use of male and female condoms as a double-barrier method is not considered acceptable due to the high failure rate when these methods are combined.

OR

-Women not of child-bearing potential may participate in the study and include those who have

* spontaneous amenorrhea for at least 12 months, not induced by a medical condition such as anorexia nervosa and not taking medications that induced amenorrhea e.g., oral contraceptives, hormones, gonadotropin-releasing hormone, anti-estrogens, selective estrogen receptor modulators, or chemotherapy; or
* spontaneous amenorrhea for 6 to 12 months and a follicle-stimulating hormone (FSH) level greater than 40 mIU/mL; or
* women with a history of hysterectomy or bilateral oophorectomy must be at least 40 years of age and FSH >40 mIU/mL.

EXCLUSION CRITERIA:

* Lifetime clinical diagnosis of schizophrenia or bipolar disorder
* BMI < 18.5 kg/m(2) and weight less than 60 Kg (both must be met)
* BMI >= 40 kg/m(2)
* History of epilepsy and/or seizures

NOTE: individuals who have a history of alcohol withdrawal seizures may be in the study as long as they have been abstinent from alcohol for at least 2 weeks prior to consent and during that period of abstinence, there were no seizure episodes (otherwise, participant remains not eligible).

* Creatinine greater than or equal to 2 mg/dL, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 times the upper normal limit, hemoglobin <10.5 g/dl
* Diagnosis of liver cirrhosis
* Clinically significant history or current eating, pituitary or adrenal gland disorders or disorder of gastric motility as judged by a study clinician as determined from medical history and/or current clinical screening information
* Current thyroid disorders that are not stable on dose of FDA-approved medications for that disease, as judged by a study clinician as determined from medical history and/or current clinical screening information. A pre-existing stable medical condition is defined as a disease not requiring significant change in therapy or hospitalization for worsening disease during the past 3 months.
* Clinically significant abnormal 12-Lead ECG
* QTcF > 450 msec for men and > 470 msec for women
* Family history of Long QT Syndrome.
* Patients on weight loss medications within 30 days of dosing
* Patients with a history of bariatric surgery
* Diagnosis of diabetes and currently on medication
* Unable to refrain from or anticipates the use of:

  * Any drugs known to be significant inhibitors of cytochrome P450 (CYP)3A enzymes and/or P-glycoprotein (P-gp) including regular consumption of grapefruit or grapefruit juice for 14 days prior to the first dose of study medication.
  * [medications like acetaminophen (up to 2 g per 24-hour period) and ibuprofen may be permitted during the study]
  * Any drugs known to be significant inducers of CYP3A enzymes and/or P-gp, including St. John's Wort, for 28 days prior to the first dose of study medication.
  * Any medications that prolong the QTcF, unless the patient has been stable on the medication for at least 3 months and has a QTcF equal to or < 450 msec
  * Benzodiazepines. If a participant received a benzodiazepine as part of their treatment during the alcohol detoxification, then s/he can still be enrolled. However, 5 half-lives (for that benzodiazepine) will be required to elapse before the anticipated date of first study drug administration
* Currently taking simvastatin >10 mg per day, atorvastatin >20 mg per day, or lovastatin >20 mg per day.

The doses of these statins in combination products should not exceed these defined dose levels.

* Patients with a history of statin-induced myopathy/rhabdomyolysis.
* Vision is unable to be corrected to (Snellen) 20/100
* Clinically-significant history of motion or car sickness, or history of vestibular disorders
* FIB-4 Score > 1.30
* Any other reason or clinical condition for which the PI or the MAI or other study clinician will consider unsafe for a possible participant to participate in this study

These criteria are based on the target population for this study. Other criteria are consistent with an ongoing study that GLWL Research Inc. is conducting with GLWL-01 in patients with Prader-Willi Syndrome (ClinicalTrials.gov NCT03274856).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.Data sharing with other protocols. Data obtained under this protocol and the National Institute on Drug Abuse (NIDA) screening protocol may be shared and combined for analysis. This will also allow us to avoid repeating assessments that are scheduled in both protocols during the same period of time, therefore avoiding duplication and minimizing participant fatigue. Participants may also consent for other NIH protocols and data collected under those protocols may be combined with data from this protocol for exploratory purposes.
  This protocol does not meet criteria for genomic data sharing. NIH Human Data Sharing (HDS) policy is not applied in this protocol because it is limited by the agreement (CRADA) with GLWL Research Inc.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Twelve months after publication
Access Criteria: To be determined.

RESULTS

PARTICIPANT FLOW:
Period: Stage I (GLWL-01 or Placebo)
Arm/Group | GLWL-01, Then Placebo | Placebo, Then GLWL-01
Started | 11 | 10
Completed | 9 | 9
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 1
Period: Washout Period
Arm/Group | GLWL-01, Then Placebo | Placebo, Then GLWL-01
Started | 9 | 9
Completed | 6 | 8
Not Completed | 3 | 1
Not completed — Physician Decision | 3 | 1
Period: Stage II (GLWL-01 or Placebo)
Arm/Group | GLWL-01, Then Placebo | Placebo, Then GLWL-01
Started | 6 | 8
Completed | 6 | 7
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were randomized to receive either GLWL-01 450 mg or placebo orally twice daily for a minimum of four days (Stage 1) followed by a minimum of two day wash-out period then cross over to receive subsequent treatment for a minimum of four days (stage II).
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with adverse events related to intervention. Adverse events were collected from participants self reporting.
Time Frame: Up to one month
Population: The analysis includes all participants who received the study interventions in each stage of the study.
Measure: Count of Participants; unit: Participants
Groups:
- GLWL-01: Participants receive GLWL-01 450 mg orally twice daily for a minimum of four days.
- Placebo: Participants receive placebo orally twice daily for a minimum of four days.
Arm/Group | GLWL-01 | Placebo
Number analyzed (Participants) | 19 | 16
Participants | 18 | 15

2. Primary Outcome: Alcohol Cue-elicited Craving Assessed in a "Bar-like" Laboratory
Description: Alcohol cue elicited craving was measured using the Alcohol Urges Questionnaire (AUQ). The AUQ is an 8-item self-administered instrument that assesses craving for alcohol among alcohol users in the current context (i.e., right now). The score ranges from 8 (lowest craving value) to 56 (highest craving value). Higher score indicated higher alcohol craving.
  AUQ was collected on each initial dosing days (2-3 days), the virtual reality buffet day (1 day), the cue-reactivity day (1 day), and the final study day (1 day), for a total of 5-6 days per intervention. The least squares average for each intervention was calculated using a linear mixed effects model including a random intercept for each participant.
Time Frame: AUQ scores were collected 5-6 days per intervention [initial dosing days (2-3 days), the virtual reality buffet day (1 day), the cue-reactivity day (1 day), and the final study day (1 day)]
Population: The analysis includes all participants who received the study interventions in each stage of the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | GLWL-01 | Placebo
Number analyzed (Participants) | 19 | 16
units on a scale | 17.8 (2.17) | 19.8 (2.19)

ADVERSE EVENTS:
Time Frame: Up to one month
Arm/Group | GLWL-01 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 18/21 | 15/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLWL-01 (N=21) | Placebo (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye movement disorder (Eye disorders) | 1 (1) | 0 (0)
Eye symptom (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 7 (7) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 2 (2)
Abnormal faeces (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (3)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (8) | 8 (10)
Hot flush (General disorders) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 3 (4)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT interval abnormal (Investigations) | 5 (6) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Oedema peripheral (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 2 (2)
Headache (Nervous system disorders) | 6 (8) | 3 (5)
Insomnia (Nervous system disorders) | 6 (7) | 5 (6)
Somnolence (Nervous system disorders) | 1 (2) | 5 (8)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Vision blurred (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 4 (4)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT03896516/Prot_SAP_000.pdf